CLINICAL TRIAL: NCT03070197
Title: Genomic Basis of Neurodevelopmental and Brain Outcomes in Congenital Heart Disease
Brief Title: Genomic Basis of Neurodevelopmental and Brain Outcomes in Congenital Heart Disease (CHD Brain and Genes)
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-6315; 5U01HL131003-02 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-01

CONDITIONS: Heart Disease Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case/CHD with deleterious mutations: Participants with CHD with damaging de novo mutations or stringently defined deleterious missense mutations) on whole exome sequencing or whole genome sequencing
  Interventions: Other: Exposure of interest: Brain MRI; Other: Exposure of interest: neurodevelopmental assessments
- Control/CHD without deleterious mutations: Participants with CHD without damaging de novo mutations or stringently defined deleterious missense mutations) on whole exome sequencing or whole genome sequencing
  Interventions: Other: Exposure of interest: Brain MRI; Other: Exposure of interest: neurodevelopmental assessments

INTERVENTIONS:
Other: Exposure of interest: Brain MRI — Brain MRI will be conducted in all participants
Other: Exposure of interest: neurodevelopmental assessments — neurodevelopmental testing will be conducted in all participants.

SUMMARY:
Approximately 400 Congenital heart disease patients will participate in the research study which will include one or more research visits for neurodevelopmental testing, brain MRI, and collection of medical history including previously collected genetic sequencing results. The investigators will explore the association between genetic variants, neurodevelopmental deficits, and brain MRI endophenotype. Analyses will compare groups with and without deleterious de novo mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in whom whole exome sequencing or whole genome sequencing has already been performed, either during the CHD GENES study or, for new centers (Utah or USCF/Stanford), after trios in existing biobanks undergo analysis by whole exome sequencing or whole genome sequencing during the Pediatric Cardiac Genomic Consortium 2 grant cycle
2. Presence of deleterious mutations (damaging de novo mutations or stringently defined deleterious missense mutations) identified on sequencing (Cases) OR absence of such known deleterious mutations (Controls)
3. Males or females, age ≥8 years
4. Diagnosis of congenital heart disease
5. Informed consent obtained

Exclusion Criteria:

1. History of cardiac transplant
2. A cardiac surgical procedure within 6 months of enrollment
3. Known clinical genetic syndrome, characterized as a monogenic condition with an identified gene associated with abnormalities of the brain structure or function, structural heart disease, and potentially other associated features.
4. Presence of CNV known to be clinically pathogenic. Variants will be classified as pathogenic using accepted types of variant evidence (e.g., population data, computational data, functional data, segregation data) as detailed in the American College of Medical Genetics and Genomics " Standards and Guidelines for the interpretation of sequence variants" (Richards et al, GIM 2015).
5. Overwhelming acquired brain injury, such as a major stroke or severe ischemic injury, that would overshadow the effect of a genetic mutation on outcome in the opinion of the center investigator
6. Lack of reading fluency in English or Spanish

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Congenital heart disease patients aged 8 years and older with prior whole exome sequencing or whole genome sequencing results
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment and behavioral health assessment | Day 1
  The investigators will compare groups with respect to achievement, IQ, learning disability, specific neuropsychological domains (e.g., memory, attention, executive functions, and visual-spatial/motor integration), adaptive function, behavior, social cognition and symptoms of autism spectrum disorder, and quality of life. The primary study outcome for this aim will be the WRAT4 composite score.

SECONDARY OUTCOMES:
Abnormalities in brain structure and microstructure on MRI | Day 1
  The investigators will compare the groups with respect to measured and derived parameters including, but not limited to, 1) regional volumetric and cortical thickness, 2) regional surface metrics, 3) voxel-based DTI eigenvectors and apparent diffusion coefficient (ADC) values, and resting state principal component analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jane Newburger, MD, Principal Investigator — Boston Children's Hospital
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Children's Hospital Boston, Boston, Massachusetts
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.benchtobassinet.org